CLINICAL TRIAL: NCT06427863
Title: Effect of Antibiotic Pretreatment on the Efficacy of WMT in the Treatment of Chronic Constipation in Adults: a Multi-center, Randomized, Placebo-controlled Clinical Study
Brief Title: Effect of Antibiotic Pretreatment on the Efficacy of WMT in the Treatment of Chronic Constipation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Faming Zhang (Other)
Responsible Party: Sponsor-Investigator, Faming Zhang, Professor, Gastroenterology, The Second Hospital of Nanjing Medical University
Organization: The Second Hospital of Nanjing Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WMT-Anti-CC-202405
Record Dates: First submitted 2024-05-20; First posted 2024-05-24 (Actual); Last update posted 2024-05-24 (Actual); Status verified 2024-05

CONDITIONS: Chronic Constipation
Keywords: chronic constipation; washed microbiota transplantation; antibiotic pretreatment; randomized controlled trial; transendoscopic enteral tube
MeSH Terms: interventions — Ornidazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Patients will receive three enemas of ornidazole 0.5g+50ml saline through the TET tube, followed by WMT once daily for a duration of 3 days.
  Interventions: Drug: Ornidazole
- Control (Placebo Comparator): Patients will receive three enemas of a placebo of equal volume through the TET tube, followed by WMT once daily for a duration of 3 days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ornidazole — Patients will receive three consecutive enemas of ornidazole 0.5g+50ml saline through the TET tube, followed by WMT treatment once daily for a duration of 3 days
  Other Names: washed microbiota transplantation
  Arms: Treatment
Drug: Placebo — Patients will receive three consecutive enemas of placebo of equal volume through the TET tube, followed by WMT treatment once daily for a duration of 3 days
  Other Names: washed microbiota transplantation
  Arms: Control

SUMMARY:
This is a randomized controlled trial to explore the efficacy of antibiotic pretreatment on the efficacy of WMT in the treatment of chronic constipation in adults: a multi-center, randomized, placebo-controlled clinical study

DETAILED DESCRIPTION:
All included in the standard but do not accord with standard of any rule out subjects will be included in this study. Demographic characteristics, complete spontaneous bowel movements（CSBM), Constipation assessment scale (CAS), Patient-Assessment of Constipation Quality Of Life（PAC-QOL) and clinical outcomes were collected. After the treatment, the efficacy and safety were evaluated during the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria to enter the study:

1. Male and female, aged ≥18 years old, provided written informed consent;
2. Subjects diagnosed with chronic constipation, with a duration of at least 6 months, and with the following conditions:

1) spontaneous bowel movement frequency <3 times/week (spontaneous bowel movement was defined as spontaneous bowel movement without rescue laxatives or manual assistance); 2) waste hard: at least 25% of defecation in Bristol stool traits scale type 1 or 2.

3. The subjects or their legal representatives gave informed consent, fully understood the purpose of the study, were able to communicate well with the researchers, and understood and complied with the requirements of the study.

Exclusion Criteria:

Subjects meeting any of the following exclusion criteria must be excluded fromthe study:

1. Presence of outlet obstruction and constipation, such as rectal mucosal prolapse
2. Combined with the results of colonoscopy in the past 24 months, those with intestinal stenosis caused by organic lesions of the digestive tract (such as tumor, inflammation, anal fissure, Crohn's disease, ulcerative colitis, intestinal adhesion, intestinal tuberculosis, etc.) and constipation;
3. Constipation caused by other systemic diseases involving the digestive tract, such as nervous system diseases (such as Parkinson's disease, spinal cord injury, multiple sclerosis, etc.), muscle diseases (such as amyloidosis, dermatomyositis, etc.), mental disorders (such as depression, etc.), metabolic and endocrine disorders (such as diabetes, hypothyroidism, etc.) or opioids, etc.
4. Has a history of abdominal pelvic surgery, but after cystic resection, cesarean section, does not appear after appendectomy postoperative intestinal complications, and intestinal polyps except after treatment;
5. Has a history of major surgery within 3 months or a history of severe trauma, and recovery is not completely;
6. There are contraindications to colonic transendoscopic intestinal tube implantation, such as severe intestinal stenosis, obstruction, deep ulcer, and high risk of operation perforation; Severe ulcers or a large number of pseudopolyps exist in the fixed area of titanium clips, which are not suitable for fixation. The subjects' behavior was seriously uncontrolled.
7. Any of the following abnormalities in cardiac function and performance:

   1. According to the New York Heart Association (NYHA) cardiac function classification, cardiac function grade Ⅲ or above;
   2. new onset myocardial infarction or unstable angina pectoris within 6 months;
   3. ECG showed QTc prolongation (QTc≥ 450ms in men and ≥470ms in women);
   4. Drug-refractory atrial arrhythmias and drug-refractory ventricular arrhythmias (including grade 2 or higher atrioventricular block).
8. Patients with poor lung function that is considered by the investigator to have an impact on the study treatment, such as patients with acute exacerbation of COPD or patients requiring long-term use of oral or intravenous steroids for control (except inhalers/sprays);
9. No control autoimmune disease and/or need long-term use of hormone (except local external use sex);
10. Patients with metabolic diseases and poorly controlled by drugs (such as thyroid dysfunction), or patients with metabolic diseases accompanied by gastrointestinal function complications (such as gastrointestinal autonomic nerve dysfunction, diabetic gastroparesis, etc.);
11. Suffering from reproductive system diseases (including but not limited to ovarian cysts, endometriosis, primary dysmenorrhea, etc.) that may lead to abdominal pain;
12. Significant laboratory abnormalities that, in the judgment of the investigator, may affect the safety of the subjects or the completion of the clinical study, including:

    A) the hemoglobin < 100 g/L; B) Serum creatinine ≥1.5 times the upper limit of normal (ULN) C) abnormal liver function, defined as AST>1.5×ULN and/or ALT>1.5×ULN and/or total bilirubin >1.5×ULN; D) blood clotting function: PLT acuities were 80 x 109 / L, APTT > 1.5 x ULN, PT > 1.5 x ULN, INR > 1.5 x ULN; E) abnormal results or defecate occult blood stool and has prompted the clinical significance of the gastrointestinal tract.
13. Have active hepatitis (requiring or taking long-term treatment), HIV, or active tuberculosis;
14. A history of drug or alcohol abuse (i.e., drinking more than 14 servings per week of beer, 45 mL of 40% spirits, or 150 mL of wine) or substance abuse;
15. The known allergic to research similar drugs, drugs or accessories;
16. Use of anti-infective drugs (antibiotics, antifungal, antiviral) within 14 days before enrollment, or need anti-infective treatment at enrollment evaluation;
17. Drugs and supplements that affect gastrointestinal motility and function cannot be stopped during the study, including but not limited to: antibiotics such as erythromycin; Drugs that modulate the intestinal microecology, such as probiotics such as Bifidobacterium; The parasympathetic nerve inhibitors, some scopolamine and atropine, belladonna, etc; Muscle relaxants, such as succinylcholine; Antidiarrheal agents such as loperamide, smecta; Opioid preparations; Drugs that inhibit gastric acid secretion;
18. Pregnant or lactating women, or refusing to use an effective contraceptive method within 3 months after the last dose of treatment;
19. 3 months prior to dosing involved in drug interventional clinical trials;
20. Suffering from malignant tumors;
21. There were other circumstances that the investigator considered inappropriate for participating in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2024-06 (Estimated); Primary Completion 2029-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Response rate of complete spontaneous bowel movements（CSBM） | One-week, Four-week and Eight-week post-WMT
  Overall CSBM respondents defined in the study of drug treatment in patients with the number of weeks of at least 50% of the time meet the CSBM weeks response week (4/8). Response was defined as a CSBM of at least three times in the week and an increase of at least one CSBM from baseline. CSBM was defined as the number of voluntary bowel movements with complete defecation sensation without taking remedial laxatives or manual assistance.
The extent of change observed in Constipation assessment scale (CAS) of participants | One-week, Four-week and Eight-week post-WMT
  The CAS consisted of 8 items, including abdominal distension, changes in exhaust volume, decreased frequency of defecation, watery stool, rectal obstruction or pressure, rectal pain during defecation, thinness of stool, and unsuccessful defecation. Each item was scored from 0 to 2 according to the severity of symptoms. Each item score was summed, with 0 as no constipation and 16 as the most severe constipation.
The extent of change observed in Patient-Assessment of Constipation Quality Of Life（PAC-QOL）of participants | One-week, Four-week and Eight-week post-WMT
  The Constipation Quality of Life Scale (PAC-QOL) contains 28 items, including physical discomfort, anxiety, psychosocial discomfort, and satisfaction. It reflects the impact of constipation on daily life in the past two weeks.

SECONDARY OUTCOMES:
The extent of change observed in stool properties of participants | One-week post-WMT
  Bristol stool form scale(BSFS) was used, which can be divided into seven types.
Rate of Adverse Events | One-week, Four-week and Eight-week post-WMT
  The rate of adverse events after antibiotic pretreatment

CONTACTS AND LOCATIONS:
Overall Officials: Faming Zhang, PhD, Principal Investigator — The Second Hospital of Nanjing Medical University
Locations (1):
- Medical Center for Digestive Diseases, The Second Affiliated Hospital of Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Keshteli AH, Millan B, Madsen KL. Pretreatment with antibiotics may enhance the efficacy of fecal microbiota transplantation in ulcerative colitis: a meta-analysis. Mucosal Immunol. 2017 Mar;10(2):565-566. doi: 10.1038/mi.2016.123. Epub 2016 Dec 21. No abstract available. PMID 28000680
- [Background] Singh P, Alm EJ, Kelley JM, Cheng V, Smith M, Kassam Z, Nee J, Iturrino J, Lembo A. Effect of antibiotic pretreatment on bacterial engraftment after Fecal Microbiota Transplant (FMT) in IBS-D. Gut Microbes. 2022 Jan-Dec;14(1):2020067. doi: 10.1080/19490976.2021.2020067. PMID 35014601
- [Background] Khalif IL, Quigley EM, Konovitch EA, Maximova ID. Alterations in the colonic flora and intestinal permeability and evidence of immune activation in chronic constipation. Dig Liver Dis. 2005 Nov;37(11):838-49. doi: 10.1016/j.dld.2005.06.008. Epub 2005 Oct 5. PMID 16169298
- [Background] Bazzocchi G, Giovannini T, Giussani C, Brigidi P, Turroni S. Effect of a new synbiotic supplement on symptoms, stool consistency, intestinal transit time and gut microbiota in patients with severe functional constipation: a pilot randomized double-blind, controlled trial. Tech Coloproctol. 2014 Oct;18(10):945-53. doi: 10.1007/s10151-014-1201-5. Epub 2014 Aug 5. PMID 25091346
- [Background] Xu J, Xu H, Guo X, Zhao H, Wang J, Li J, He J, Huang H, Huang C, Zhao C, Li Y, Zhou Y, Peng Y, Nie Y. Pretreatment with an antibiotics cocktail enhances the protective effect of probiotics by regulating SCFA metabolism and Th1/Th2/Th17 cell immune responses. BMC Microbiol. 2024 Mar 18;24(1):91. doi: 10.1186/s12866-024-03251-2. PMID 38500062